CLINICAL TRIAL: NCT04325841
Title: Phase II Study of Autologous Murine Anti-CD19 Chimeric Antigen Receptor T Cells Treating Refractory or Relapsed B Acute Lymphoblastic Leukemia Children
Brief Title: Phase II Study of Anti-CD19 CAR-T Cells Treating Leukemia Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Boren Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BR-19-C
Record Dates: First submitted 2020-03-26; First posted 2020-03-30 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Acute Lymphoblastic Leukemia, Pediatric; Acute Lymphoblastic Leukemia, in Relapse; Refractory Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Autologous Murine Anti-CD19 CAR-T treatment (Experimental)
  Interventions: Biological: Murine autologous anti-CD19 chimeric antigen receptor T cells

INTERVENTIONS:
Biological: Murine autologous anti-CD19 chimeric antigen receptor T cells — CAR-T cells were manufactured from peripheral blood mononuclear cells collected by leukapheresis and frozen for multiple uses. Before each CAR T-cell infusion (day 0), patients received lymphodepleting chemotherapy composing of Fludarabine (30 mg/m2/day) and Cyclophosphamide (250 mg/m2/day) on days -5 to -3. No bridging chemotherapy was given between enrollment and infusion. In CD19 T cell clinical trials, CAR-T cells was given once. All patients underwent bone marrow (BM) biopsy examination and radiology studies on days 30 and every month to determine the response and remission status. Bone biopsy, MRD status by FCM and RT-PCR (if the patient had fusion gene), and EMDs evaluation by CT/MRI/PET-CT were also conducted before CAR-T cell infusion to determine the disease status.

SUMMARY:
The investigators will conduct a phase II clinical trial of autologous murine anti-CD19 chimeric antigen receptor T cells treating refractory or relapsed B acute lymphoblastic leukemia children in Beijing Boren Hospital. The study will be approved by the institutional review board of Beijing Boren Hospital, and informed consent will be obtained in accordance with the Declaration of Helsinki. All these participants will be matched the diagnostic criteria for (r/r) B-ALL according to the WHO classiﬁcation and complete morphological evaluation, immunophenotype analysis by flow cytometry (FCM), cytogenetic analysis by routine G-banding karyotype analysis and leukemia fusion gene screening by multiplex nested reverse transcriptase-polymerase chain reaction (PCR). Participants will be eligible if they are heavily treated B-ALL who failed from re-induction chemotherapy after relapse or continued MRD+ for more than three months, and had positive CD19 expression on leukemia blasts by FCM (>95% CD19). After CAR T-cell infusion, clinical outcomes including overall survival (OS), Disease-free survival (DFS), adverse effects and relapse will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were diagnosed as primary refractory or relapsed B-ALL. All the patients matched the diagnostic criteria of ALL according to the WHO classification and conducted morphological evaluation, immunophenotype analysis by flow cytometry (FCM), cytogenetic analysis by routine G-banding karyotype analysis, screen of 56 leukemia-related fusion genes by multiplex nested reverse transcriptase-polymerase chain reaction (RT-PCR), and quantification of fusion genes by real-time PCR with ABL1 as reference. Extramedullary diseases (EMDs) were confirmed CD19+ by FCM and evaluated by positron emission tomography/computed tomography (PET/CT), CT, MRI or ultrasonography. The patient relapsed during chemotherapy or failed from re-induction chemotherapy (including first and second-generation TKIs) after relapse or had a persistent positive minimal residual disease (MRD) for three months. Patients had positive CD19 expression on leukemia blasts by FCM (>95% CD19 positive);
* Age from 0 to 18 years old;
* Children candidates can be recruited after the legal guardian or patient advocate has signed the treatment consent form and voluntary consent form;

Exclusion Criteria:

* Intracranial hypertension or unconscious;
* Acute heart failure or severe arrhythmia;
* Acute respiratory failure;
* Other types of malignant tumors;
* Diffuse intravascular coagulation;
* Serum creatinine and/or blood urea nitrogen over 1.5 times than normal range;
* Sepsis or other uncontrolled infection;
* Uncontrolled diabetes mellitus;
* Severe psychological disorder;
* Obvious cranial lesions with cranial MRI;
* More than 20 counts/ul leukemic cells in cerebrospinal fluid;
* More than 30% leukemic cells in the blood;
* Stage III WHO/ECOG score;
* Organ recipients;
* Pregnant or breastfeeding;
* Active, uncontrolled infection, including hepatitis B, hepatitis C or human immunodeficiency virus (HIV);

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2022-03-24 (Actual); Primary Completion 2024-04-03 (Actual); Study Completion 2024-04-03 (Actual)

PRIMARY OUTCOMES:
CR rate | 1 month
  The complete remission(CR) rate to the CAR-T treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Boren Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No